CLINICAL TRIAL: NCT02563808
Title: Impact of Anticipated Regret on Decision-Making in Preference Sensitive Care for Breast and Prostate Cancer
Brief Title: Impact of Anticipated Regret Incorporation Into Patient Decision Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 817436
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Regret

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Decision Aid (Active Comparator): The brochure with standard information on surgery for early-stage breast cancer
  Interventions: Other: Standard Decision Aid
- Post-surgical Regret Decision Aid (Experimental): The brochure that incorporates additional information on the rates of regret after surgical treatment of early-stage breast cancer.
  Interventions: Other: Post-surgical Regret Decision Aid

INTERVENTIONS:
Other: Standard Decision Aid — Females will receive standard decisions aid for early stage breast cancer.
  Arms: Standard Decision Aid
Other: Post-surgical Regret Decision Aid — Females will receive anticipated regret-augmented version for early breast cancer.
  Arms: Post-surgical Regret Decision Aid

SUMMARY:
The purpose of this study is to investigate the impact of incorporating "anticipated regret " into standard patient decision aids. Participants in the Wharton Behavioral Lab will be administered a standard patient decision aid and an "anticipated regret" augmented decision aid. Participants will complete a computerized survey about their experiences with each version, and their answers will be assessed for potential differences associated with the incorporation of "Anticipated Regret."

DETAILED DESCRIPTION:
Participants will be recruited through the Wharton Behavioral Lab. Upon arrival males will be provided with two decision aids focusing on prostate cancer, while females will be provided with two decision aids focusing on early breast cancer. One of these decision aids will be a standard version, and one of these will be the anticipated regret-augmented version. Participants will be randomized to which version they receive first to minimize the effect of presentation order. After reviewing the materials, participants will immediately complete a computerized survey at their work stations that will ask them to answer questions based on the materials presented as well as how any hypothetical treatment decisions they would be asked to make would have been influenced by them. Because these are healthy subjects participating in a hypothetical decision-making process for sole purpose of research, the intervention can neither be categorized as experimental or as the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females ages 18 years or older

Exclusion Criteria:

* Under age 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy females ages 18 and older
Enrollment: 189 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Fleisher, MD, Principal Investigator — UPenn, Chairman, Anesthesiology & Critical Care

REFERENCES:
- [Derived] Speck RM, Neuman MD, Resnick KS, Mellers BA, Fleisher LA. Anticipated regret in shared decision-making: a randomized experimental study. Perioper Med (Lond). 2016 Mar 2;5:5. doi: 10.1186/s13741-016-0031-6. eCollection 2016. PMID 26941952

RESULTS

PARTICIPANT FLOW:
Groups:
- Survey: Standard Version: Females will receive standard decisions aid for early stage breast cancer.
  Survey: Standard
- Survey: Anticipated Regret Version: Females will receive anticipated regret-augmented version for early breast cancer.
  Survey: Regret
Period: Overall Study
Arm/Group | Survey: Standard Version | Survey: Anticipated Regret Version
Started (A total of 5 participants enrolled were not included in final data due to data collection error) | 96 | 88 (A total of 5 participants enrolled were not included in final data due to data collection error)
Completed | 96 | 88
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two participants did not complete the demographic questions. As such only 94 are being analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Survey: Standard Version | Survey: Anticipated Regret Version | Total
Number analyzed (Participants) | 94 | 88 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 88 | 182
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (7.2) | 21.8 (5.9) | 22.0 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Female only
  Participants
    Female | 94 | 88 | 182
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 82 | 72 | 154
  Unknown or Not Reported | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 33 | 35 | 68
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 13 | 32
  White | 30 | 24 | 54
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 94 | 88 | 182

OUTCOME MEASURES:

1. Primary Outcome: Difference in Consideration of Regret
Description: Compare decisions about a hypothetical surgery for breast cancer, and examined whether regret is a consideration in treatment decisions between those who received the experimental and those who received the standard version of the decision aid. The values represent numbers of participants who reported that regret played a role in their decision-making.
Time Frame: 11 months
Measure: Number; unit: participants reported regret played role
Arm/Group | Survey: Standard Version | Survey: Anticipated Regret Version
Number analyzed (Participants) | 96 | 88
participants reported regret played role | 62 | 69

ADVERSE EVENTS:
Arm/Group | Survey: Standard Version | Survey: Anticipated Regret Version
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/88
Other Adverse Events (participants affected / at risk) | 0/94 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes